CLINICAL TRIAL: NCT00312260
Title: Randomized Controlled Trial Comparing Gabapentin and Amitriptyline for the Treatment of Neuropathic Pain in Children and Adolescents
Brief Title: Comparing Gabapentin and Amitriptyline for the Treatment of Neuropathic Pain in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Stephen Brown, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000008259
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pain
Keywords: Pain; Analgesia; Gabapentin; Amitriptyline; Pediatrics
MeSH Terms: conditions — Pain; Agnosia | interventions — Gabapentin; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Gabapentin
- 2 (Active Comparator)
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Gabapentin — Gabapentin will be prescribed at 900mg/d (300mg tid). A dose escalation schedule will be followed: one pill taken at night (~2000h) for the first 3 days, one pill at night and one pill in the morning (~0800h) for the second 3 days and finally, one pill at night, one in the morning and one mid-afternoon (~1400h) for the reminder of the trial.
  Arms: 1
Drug: Amitriptyline — Amitriptyline will be prescribed at a dose of 10mg (qhs). A dose escalation schedule will be followed: one pill taken at night (~2000h) for the first 3 days, one pill at night and one pill in the morning (~0800h) for the second 3 days and finally, one pill at night, one in the morning and one mid-afternoon (~1400h) for the reminder of the trial.
  Arms: 2

SUMMARY:
The objective of the study is to compare the efficacy of gabapentin and amitriptyline for treating neuropathic pain in children in a randomized controlled trial.

DETAILED DESCRIPTION:
Clinical experience and case reports suggest that both amitriptyline and gabapentin are effective treatments for neuropathic pain in children; however we do not know which drug is more effective for specific pain conditions or for specific children. This study will be the first prospective, randomized double-blind controlled trial directly comparing gabapentin and amitriptyline for the treatment of neuropathic pain in a paediatric population. We will also study the time course for pain reduction and evaluate changes in children's physical function, mood, and sleep. This information is needed to determine which drug is better for which children and which pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* 8 - 17 years of age
* Diagnosis of neuropathic pain

Exclusion Criteria:

* Additional health problems
* Lactose intolerant
* Unable to swallow size 0 gelatin capsules
* Pregnant
* Unable to speak English

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2010-05 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
change in child's pain intensity score | 6 weeks

SECONDARY OUTCOMES:
change in child's pain-related disability ratings | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Brown, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada